CLINICAL TRIAL: NCT05583370
Title: The Effect of Aflatoxin Metabolites Concentration in Follicular Fluid on Laboratory and Clinical Outcomes in Intracytoplasmic Sperm Injection Cycles
Brief Title: The Effect of Aflatoxin Metabolites Concentration in Follicular Fluid on Laboratory and Clinical Outcomes in ICSI
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Romany Hany, Principal investigator, Assiut University
Other Study IDs: Aflatoxins effect in ICSI
Record Dates: First submitted 2022-10-10; First posted 2022-10-17 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Aflatoxin Poisoning
Keywords: Aflatoxins and ICSI
MeSH Terms: conditions — Aflatoxin Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mycotoxins are secondary toxic metabolites produced by Aspergillus, Penicillium, and Fusarium species of fungi, when they infect and proliferate on various agricultural commodities either in the field and/or during storage. The well-known detrimental health effects of mycotoxins in humans include liver cancer, Balkan endemic nephropathy, child growth impairment, immune suppression, neural tube defects and death in acute exposure. However, growing evidence also suggests that mycotoxins may negatively influence human fertility.

DETAILED DESCRIPTION:
Aflatoxins (AFs) contaminate different types of food and feed commodities, especially in hot and humid regions of the world . The major AFs are characterized as B1, B2, G1 and G2, among these four, B1 is best known because of its hepatocarcinogenic nature ]. AFs M1 and M2 are produced by biological metabolism of AFB1 and AFB2 from contaminated feed used by animals and excreted in milk and dairy products.

Natural occurrence of mycotoxins is present in a large part of the world food supply and bear potential threat to food safety and food security . From global perspective of food safety and food security, mycotoxins contamination of foods has gained much attention as potential health hazards for humans and animals.

Studies using animal and cell models indicate that zearalenone, deoxynivalenol, ochratoxin A and aflatoxin B1 can adversely affect fertility, mainly through damage to sex organs, gametes and disruption of steroidogenesis. For instance, animal models have indicated that exposure to the aforementioned mycotoxins can promote adverse effects on spermatozoa, sertoli and Leydig cell function, oocyte maturation, and uterine and ovarian development and function, both in vivo and ex vivo. They may also induce oxidative stress resulting in sperm DNA damage and subsequently, reduced fertilisation rates and lower embryo quality. Furthermore, mycotoxins may act as endocrine disrupters, altering the steroid hormone homeostasis, consequently leading to subfertility or infertility. In humans, zearalenone has been linked to precocious puberty in girls, correlating with extremely high serum oestrogen levels whereas aflatoxin B1 has been linked to poor sperm quality in infertile males. Considering that multiple exposures to these mycotoxins have been reported in humans and that there is a homology in organ systems between animals and humans, these findings may have clinical relevance in human infertility.

ELIGIBILITY:
1. Inclusion criteria:

   * Infertile women undergoing in vitro fertilization with intracytoplasmic sperm injection (IVF/ICSI) and fresh embryo transfer at the Unit aged between 18 and 39 years
   * Indications for IVF will be either ovulatory disorders, tubal disorders, or unexplained infertility.
   * All down-regulation protocols and all types of gonadotropins for ovarian stimulation will be included.
2. Exclusion criteria:

   * Patients who refuse to participate in clinical research
   * Significant medical disease (hypertension, diabetes mellitus, cardiac disease, blood disease, etc.)
   * Male factor infertility.
   * Women with confirmed intrauterine lesions, i.e. polyps, submucous myomas, adhesions, septa or hydrosalpinges. Women with these lesions will be only included if corrected.
   * Women with expected poor response to ovarian stimulation; defined as antral follicle count less than 5, anti-mullerian hormone (AMH) less than 0.8 ng/mL or a history of previous IVF cycle that yielded less than 5 oocytes.
   * Women undergoing IVF not ICSI as the method of insemination for all retrieved oocytes.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing IVF with ICSI as the method of insemination
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
- Clinical pregnancy | 4 weeks from embryo transfer
  - Clinical pregnancy: the presence of gestational sac and fetal pole with visible pulsations after 4 weeks from embryo transfer.

SECONDARY OUTCOMES:
Biochemical pregnancy | 2weeks from embryo transfer
  positive bHCG in the serum measured 2 weeks after embryo transfer
Oocyte quality | Immediately after ovum pick up
  Percentage of good quality oocytes: the number of good quality oocytes divided by the total number of retrieved oocytes x 100
Fertilization rate | 16-18 hours after insimination
  the number of fertilized oocytes divided by the total number of injected oocytes x 100
Embryo quality | 3-5 days after ovum pick up
  - Percentage of good-quality embryos: the number of good-quality embryos divided by the total number of injected oocytes x 100 assessed on the day of embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Romany H Gerges, Resident, Principal Investigator — Assiut University
Locations (1):
- Assiu University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided